CLINICAL TRIAL: NCT04639986
Title: A Phase 3 Asian Study of Sacituzumab Govitecan (IMMU-132) Versus Treatment of Physician's Choice (TPC) in Subjects With Hormonal Receptor-positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Metastatic Breast Cancer (MBC) Who Have Failed at Least 2 Prior Chemotherapy Regimens
Brief Title: Asian Study of Sacituzumab Govitecan (IMMU-132) in HR+/HER2- Metastatic Breast Cancer (MBC)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVER-132-002; CTR20210096 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform)
Record Dates: First submitted 2020-11-17; First posted 2020-11-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Breast Cancer
Keywords: sacituzumab govitecan; IMMU-132; Unresectable or Metastatic Breast Cancer; hormonal receptor; HR positive; Anti-TROP2; Human epidermal growth factor receptor 2 (HER2) Negative; Antibody Drug Conjugate
MeSH Terms: conditions — Breast Neoplasms | interventions — sacituzumab govitecan; eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan-hziy (Experimental): Participants will receive Sacituzumab Govitecan-hziy 10 mg/kg on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive recommended doses and schedules as per package insert depending on region.
  * Eribulin (1.4 mg/m^2 of eribulin mesylate or 1.23 mg/m^2 of eribulin on Days 1 and 8 of a 21-day cycle)
  * Capecitabine (1000 to 1250 mg/m^2 twice daily on Days 1 to 14 of a 21-day cycle)
  * Gemcitabine (800 to 1200 mg/m^2 on Days 1, 8, and 15 of a 28-day cycle)
  * Vinorelbine (25 mg/m^2 on Day 1 weekly)
  Interventions: Drug: Eribulin Mesylate Injection; Drug: Capecitabine Oral Product; Drug: Gemcitabine Injection; Drug: Vinorelbine injection

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Sacituzumab govitecan 10 mg/kg via IV injection administered on Days 1 and 8 of a 21-day cycle. Subjects will continue to receive study treatment until PD as judged by local investigator review, development of unacceptable toxicity, or withdrawal of consent.
  Other Names: IMMU-132; Trodelvy™; GS-0132
  Arms: Sacituzumab Govitecan-hziy
Drug: Eribulin Mesylate Injection — Eribulin is administered by intravenous (IV) following recommended doses and regimens as per approved package inserts.
  Other Names: Halaven
  Arms: Treatment of Physician's Choice (TPC)
Drug: Capecitabine Oral Product — Capecitabine is administered orally (PO) following recommended doses and regimens as per approved package inserts.
  Other Names: Xeloda
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine Injection — Gemcitabine is administered by intravenous (IV) following recommended doses and regimens as per approved package inserts.
  Other Names: Gemzar
  Arms: Treatment of Physician's Choice (TPC)
Drug: Vinorelbine injection — Vinorelbine is administered by intravenous (IV) following recommended doses and regimens as per approved package inserts.
  Other Names: Navelbine
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The goal of this study is to compare the study drug, sacituzumab govitecan-hziy, versus doctors' treatment of choice in participants with HR+/HER2- metastatic breast cancer (MBC) who have failed at least 2 prior chemotherapy regimens.

DETAILED DESCRIPTION:
Approximately 330 eligible participants will be randomly allocated to one of the following 2 treatment arms in a 1:1 ratio:

Investigational Arm:

Sacituzumab Govitecan-hziy 10 mg/kg via intravenous (IV) injection administered on Day 1 and Day 8 (21-day cycle).

Control Arm:

Recommended doses and schedules as per package insert depending on region. Eribulin; Capecitabine; Gemcitabine; Vinorelbine Participants will be treated until disease progression as judged by local investigator review, development of unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Key Inclusion Criteria:

* Female or male individuals aged ≥18 years at the time of signing the informed consent form
* Documented evidence of hormone receptor-positive HER2-negative (HR+/HER2-) MBC confirmed
* Refractory to or relapsed after at least 2, and no more than 4, prior systemic chemotherapy regimens for MBC
* Should have been previously treated with at least 1 taxane in any setting, at least 1 prior anticancer hormonal treatment in any setting
* Eligible for one of the chemotherapy options listed in the TPC arm
* Documented radiographic disease progression after the most recent therapy
* Measurable disease by CT or MRI in accordance with RECIST v 1.1, bone-only disease is not measurable and is not permitted.
* Adequate bone marrow function, hepatic and renal function
* Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta human chorionic gonadotropin [ß-hCG]

Key Exclusion Criteria:

* Previous treatment with Topoisomerase 1 Inhibitors as a free form or as other formulations
* Individuals who have known brain metastases.
* Have an active second malignancy within 3 years prior to providing informed consent
* Individuals with active hepatitis B virus (HBV), or hepatitis C virus infection (measurable viral RNA load with polymerase chain reaction).
* Active serious infection requiring systemic antibiotic use within 7 days before Cycle1 Day 1.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Known hypersensitivity or intolerance to either of the study treatments or any of the excipients.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 4 years
  PFS is defined as from the date of randomization until the date of disease progression (PD) or death, whichever occurs earlier. Disease progression will be determined according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1) by Independent Reviewing Committee (IRC).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 4 years
  OS is defined as from the date of randomization to death from any cause.
Objective Response Rate (ORR) by IRC | Up to 4 years
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR).
Duration of Response (DOR) by IRC | Up to 4 years
  DOR is defined as from the date of first onset of tumor response (CR or PR) to PD or death, whichever occurs earlier.
Clinical Benefit Rate (CBR) by IRC | Up to 4 years
  CBR is defined as best overall response of CR or PR or durable stable disease (SD) (duration of SD ≥ 6 months after randomization).
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | First dose date up to 4 years plus 30 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) According to NCI CTCAE Version 5.0 | First dose date up to 4 years plus 30 days
Change From Baseline of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire, Core 30, Version 3.0 (EORTC QLQ-C30) Score | Baseline, up to 4 years
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) to assess 15 scales; 1 global health status/quality of life (QOL), 5 functional scales (physical, role, cognitive, emotional, and social), and 9 symptom/item scales(fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of function, a high score for the global health status/QOL represents a high QOL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change From Baseline of the European Quality of Life 5-Dimensions 5 Levels Instrument (EuroQOL EQ-5D-5L) Score | Baseline, up to 4 years
  The EQ-5D-5L is an instrument for use as a measure of health outcome.The EQ-5D-5L consists of 2 sections: the EuroQoL (5 dimensions) (EQ-5D) descriptive system and the EuroQoL visual analogue scale (EQ-VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ-VAS indicate better health.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events Assessed by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (NCI PRO-CTCAE) | Baseline, up to 4 years
  NCI PRO-CTCAE is a patient-reported item library used to evaluate symptomatic treatment-emergent adverse events in participants on cancer clinical trials. The items selected for this study include: decreased appetite, nausea, vomiting, constipation, diarrhea, abdominal pain, shortness of breath, hair loss, and fatigue.
Pharmacokinetic (PK) Parameter: Cmax of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Tmax of of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Tmax is defined as the time to maximum drug concentration.
PK Parameter: Ctrough of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Ctrough is defined as the concentration of drug at the end of the dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (43):
- China (27):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - The First Hospital of Jilin University, Changchun
  - Chongqing University Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat Sen Memorial Hospital of Sun Yat sen University, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Sir Run run Shaw hospital Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The second Hospital of Anhui Medical University, Hefei
  - Shandong Cancer Hospital, Jinan
  - Yunnan Cancer Hospital, Kunming
  - Linyi Cancer Hospital, Linyi
  - Jiangsu Province Hospital, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai General Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- South Korea (8):
  - Dong-A University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (8):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu B, Wang S, Yan M, Sohn J, Li W, Tang J, Wang X, Wang Y, Im SA, Jiang D, Valdez T, Dasgupta A, Zhang Y, Yan Y, Komatsubara KM, Chung WP, Ma F, Dai MS. Sacituzumab govitecan in HR+HER2- metastatic breast cancer: the randomized phase 3 EVER-132-002 trial. Nat Med. 2024 Dec;30(12):3709-3716. doi: 10.1038/s41591-024-03269-z. Epub 2024 Oct 1. PMID 39354196
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04639986